CLINICAL TRIAL: NCT05381519
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of DXP604 in Patients With Mild to Moderate COVID-19
Brief Title: A Study to Evaluate the Efficacy and Safety of DXP604 in Patients With Mild to Moderate COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DXP604-201
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — DXP-604

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DXP604 (Experimental): 1800mg，IVgtt
  Interventions: Biological: DXP604
- placebo (Placebo Comparator): IVgtt
  Interventions: Biological: DXP604

INTERVENTIONS:
Biological: DXP604 — 1800mg，IVgtt

SUMMARY:
A phase II, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of DXP604 in patients with mild to moderate COVID-19.

By determination of severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) virus in nasopharyngeal swab samples by reverse transcription quantitative polymerase chain reaction (RT-qPCR) from baseline (2 h ± 30 min before dosing) to Viral load changes on day 8,to evaluate the efficacy of DXP604 monotherapy in patients with mild to moderate coronavirus disease 2019 (COVID-19).

It was assumed that the difference in viral load change of SARS-CoV-2 virus from baseline (2 h ± 30 min before administration) to day 8 in nasopharyngeal swab samples by RT-qPCR between the experimental drug group and the placebo group was -1.00 log10 copies/mL.The null and alternative hypotheses comparing the experimental drug group with the placebo group are set as follows:

H0：µ1 = µ2 H1：µ1 ≠ µ2

ELIGIBILITY:
Inclusion Criteria:

1. The age of the subjects when signing the ICF is 18 to 70 years old (including 18 and 70 years old), male or female;
2. Possess venous access conditions, allowing drug administration and blood sample collection according to the research protocol;
3. SARS-CoV-2 positive in any laboratory-confirmed sample within 96 hours before screening;
4. According to the National Health Commission of the People's Republic of China (NHC) "New Coronary Virus Pneumonia Diagnosis and Treatment Program", the ninth revised version of the trial was clinically classified as mild/ordinary patients;
5. There is at least one factor that may lead to a high risk of severe/critical COVID-19: ① age > 60 years; ② cardiovascular and cerebrovascular diseases (including hypertension), chronic lung diseases (chronic obstructive pulmonary disease, chronic obstructive pulmonary disease, Moderate to severe asthma), diabetes, chronic liver, kidney disease, tumor and other basic diseases; ③ immunodeficiency (such as AIDS patients, long-term use of corticosteroids or other immunosuppressive drugs lead to immunosuppression); ④ obesity (physical constitution) index ≥ 30); ⑤ Heavy smokers.
6. Symptoms of COVID-19 ≤ 5 days before randomization; such as fever, cough, shortness of breath, sore throat, diarrhea, vomiting, and dysgeusia;
7. Agree to collect nasopharyngeal swabs, saliva and venous blood;
8. The subjects can communicate well with the researcher, understand and comply with the requirements of this study, and understand and sign the ICF.

Exclusion Criteria:

1. Severe COVID-19 patients who meet any of the following:

   * Shortness of breath, respiratory rate ≥ 30 times/min;
   * In resting state, blood oxygen saturation (SpO2) ≤ 93% when inhaling air;
   * Arterial blood oxygen partial pressure PaO2/inhaled oxygen concentration (FiO2)≤300mmHg (1mmHg=0.133kPa); Note: For areas with high altitude (over 1000 meters above sea level), the following formula should be used to correct PaO2/FiO2: PaO2/FiO2×[760/air pressure (mmHg)];
   * The clinical symptoms are progressively worsened, and lung imaging shows that the lesion progresses significantly within 24 to 48 hours by >50%;
2. Critically ill patients with COVID-19 who meet any of the following:

   * Respiratory failure occurs and requires mechanical ventilation;
   * Shock occurs;
   * Complicated with other organ failure requires ICU monitoring and treatment;
3. Those who are known to be allergic to the test drug and its components;
4. Hemodynamic instability within 24 hours before treatment allocation requires the use of vasopressors;
5. Suspected or confirmed serious, active bacterial, fungal, viral or other infections (except for COVID-19) that the investigator believes may pose a risk when taking interventions;
6. Any comorbidities requiring surgery within 7 days prior to screening, or comorbidities deemed life-threatening within 29 days prior to screening;
7. Any serious concomitant systemic disease, condition or disorder that the investigator believes should be prevented from participating in this study;
8. Patients with positive anti-SARS-CoV-2 immunoglobulin G (IgG) and IgG>10;
9. Patients with malignant tumors who are undergoing chemotherapy and radiotherapy before and after surgery;
10. Those who have received SARS-CoV-2 specific immunoglobulin (including monoclonal antibody) therapy;
11. Those who have completed the vaccination against COVID-19 within 1 month;
12. Those who have a history of receiving convalescent COVID-19 plasma treatment;
13. Received any study treatment for COVID-19 within 30 days prior to administration, including but not limited to antiviral drugs, corticosteroids, interleukin-1 inhibitors, interleukin-6 inhibitors, and intravenous immunoglobulin;
14. Participated in clinical trials of other drugs within 3 months before screening;
15. Those who are dizzy with acupuncture and blood;
16. Within 4 months after signing the ICF to the end of the trial, those who have a childbearing plan or who do not agree to take effective non-drug contraceptive measures during this period;
17. Pregnant and lactating women;
18. Other factors considered by the investigator to be inappropriate for entry into this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
viral load of SARS-CoV-2 virus in nasopharyngeal swab samples | from baseline (2 h ± 30 min before dosing) to day 8
  determination of changes in viral load of SARS-CoV-2 virus in nasopharyngeal swab samples from baseline (2 h ± 30 min before dosing) to day 8

IPD SHARING:
Plan to Share IPD: No